CLINICAL TRIAL: NCT01337661
Title: An Exploratory Study of the Cellular Inflammatory Mechanisms Associated With Chronic Obstructive Pulmonary Disease Exacerbations
Brief Title: A Study of the Inflammatory Pathways Associated With Chronic Obstructive Pulmonary Disease Exacerbations
Status: Completed | Type: Observational
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CD-RI-INDP-1048
Record Dates: First submitted 2011-04-13; First posted 2011-04-19 (Estimated); Last update posted 2012-08-28 (Estimated); Status verified 2012-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease; COPD; Acute Exacerbation of COPD; AECOPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood, Endobronchial tissues and Bronchoalveolar (BAL) samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- COPD subjects: Adult male and female subjects with COPD

SUMMARY:
The purpose of this study is to observe how the inflammatory pathways differ in subjects with chronic obstructive pulmonary disease (COPD) during an acute exacerbation of COPD (AECOPD).

DETAILED DESCRIPTION:
This is an observational study in adult male and female subjects with COPD to collect blood, endobronchial tissues and BAL to investigate the inflammatory genes/pathways associated with AECOPD at the time of exacerbation (ie, active disease) and at 6 weeks later (ie, stable disease).

ELIGIBILITY:
Inclusion Criteria:

* Physician-diagnosed acute exacerbations of chronic obstructive pulmonary disease
* Current or ex-smoker with a tobacco history of 15 or more pack years
* Females of childbearing potential must use birth control for the duration of the study.

Exclusion Criteria:

* Evidence or history of clinically significant disease
* Subjects with asthma
* Subjects taking anti-leukotriene medications

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects referred to the hospital clinic with AECOPD
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2011-04; Primary Completion 2012-01 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Identification of how inflammatory pathways differ in COPD subjects | 6 weeks
  Identify how inflammatory pathways differ in subjects with COPD during an acute exacerbation relative to when the disease is stable.

SECONDARY OUTCOMES:
Biomarker Sample Repository | 6 weeks
  Establish a biomarker sample repository to support future target validation for the treatment of subjects with COPD.

CONTACTS AND LOCATIONS:
Overall Officials: Rene van der Merwe, MBChB, MFPM, Study Director — MedImmune Ltd; Prof. Connor Burke, Principal Investigator — BCF Diagnostics
Locations (1):
- Research Site, Dublin, Ireland